CLINICAL TRIAL: NCT07274800
Title: Adjuvant Ultra Hypofractionation Radiotherapy Versus Hypofractionation Radiotherapy in Treatment of Early Invasive Breast Cancer
Brief Title: Adjuvant Ultra-Hypofractionated vs Hypofractionated Radiotherapy for Early Breast Cancer
Acronym: UHF vs HF-EBC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11119
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A:Adjuvat Ultra-Hypofractionation Radiotherapy (Experimental): Adjuvant external beam radiotherapy after breast-conserving surgery Total dose: 26 Gy delivered in 5 fractions over 1 week 3D conformal radiotherapy technique without breath-hold Daily fractionation, whole breast irradiation
  Interventions: Radiation: Adjuvant Ultra hypofractionation radiotherapy
- Arm B: Adjuvant hypofractionation radiotherapy (Experimental)
  Interventions: Radiation: Adjuvant Hypofarctionated radiotherapy

INTERVENTIONS:
Radiation: Adjuvant Ultra hypofractionation radiotherapy — Adjuvant external beam radiotherapy after breast-conserving surgery Total dose: 26 Gy delivered in 5 fractions over 1 week 3D conformal radiotherapy technique without breath-hold Daily fractionation, whole breast irradiation
  Arms: Arm A:Adjuvat Ultra-Hypofractionation Radiotherapy
Radiation: Adjuvant Hypofarctionated radiotherapy — Adjuvant external beam radiotherapy after breast-conserving surgery Total dose: 40 Gy delivered in 15 fractions over 3 week 3D conformal radiotherapy technique without breath-hold Daily fractionation, whole breast irradiation
  Arms: Arm B: Adjuvant hypofractionation radiotherapy

SUMMARY:
breast-conserving surgery. One group receives ultra-hypofractionated radiotherapy (26 Gy in 5 sessions over 1 week), while the other group receives hypofractionated radiotherapy (40 Gy in 15 sessions over 3 weeks). The study aims to compare skin toxicity, cosmetic outcomes, and local cancer control between thetwo schedules . Participants are followed during and after radiotherapy for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:• Histological diagnosis of breast adenocarcinoma

* Prior breast conservative surgery negative resection margins (3 mm)
* Pathological stage pT1-pT2, N0-1, pT3-N0, M0
* No macroscopic evidence of distant metastases at diagnosis
* Age 18-80 years
* Female patients
* Normal hematological and biochemical laboratory tests
* Written informed consent was obtained from all patients

Exclusion Criteria: • Patients underwent mastectomy.

* Locally advanced disease pT4, N2,3.
* Positive surgical margins
* Prior thoracic radiation
* Synchronous second primary tumor
* Distant metastases
* Pregnancy
* Presence of a concomitant psychiatric disorder precluding an aware informed consent.
* Age >80 years
* Low risk patient meeting all the following criteria (more than or equal 65 years, PT1, grade 1 or 2, +ER, -Her2nu, N0, M0).

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2025-11-27 (Actual); Study Completion 2025-11-27 (Actual)

PRIMARY OUTCOMES:
Acute Skin Toxicity (CTCAE v5.0) | From start of radiotherapy to 6 weeks post-treatment
  Incidence and severity of acute skin toxicity (erythema, desquamation, edema) assessed

SECONDARY OUTCOMES:
Late Skin Toxicity and Cosmesis | 12 months post-radiotherapy
  Incidence of late skin changes (pigmentation, fibrosis) and cosmetic outcomes assessed at 12 months post-radiotherapy using physician assessment and patient-reported outcomes (EORTC QLQ)
Locoregional Recurrence | Up to 24 months post-radiotherapy
  Rate of locoregional recurrence in the irradiated breast assessed by clinical examination and imaging at follow-up visits

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig University, Zagazig, Egypt